CLINICAL TRIAL: NCT06535126
Title: Safety and Tolerability Studies of CanProFem-AK, Vaginal Suppositories in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Industrial Microbiology LLP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ПМ-002-23г
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Candidosis Vaginal
Keywords: phase I of clinical trial; Candida; antifungal drug; antibiotic; suppository
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Torulopsis

STUDY DESIGN:
Intervention Model Description: Objectives of the study: Determine the safety and tolerability of CanProFem-AK, 100 mg suppositories in healthy volunteers.
  The study includes the following stages:
  Stage 1 of the study (introductory stage) included recruitment and screening of healthy volunteers - study participants, signing of informed consent, medical examination and laboratory tests.
  Stage 2 of the study (baseline control stage) involved clinical measurements taken before the start of the study (baseline measurements) for each subject. These measurements were conducted to obtain baseline data, which were then compared with the results obtained after the study's conclusion.
  Stage 3 of the study included medical observation after the vaginal administration of one suppository, including gynecological examination and bacterial culture sampling from the vagina at 3, 6, 9, 12, and 24 hours. Additional blood and urine tests will be performed after 24 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): The drug administration scheme involves vaginal administration of one suppository (CanProFem-AK, 100 mg). The total duration of participation in a study is one day.
  Interventions: Drug: CanProFem-AK

INTERVENTIONS:
Drug: CanProFem-AK — Dosage form - vaginal suppositories (100 mg). Dosage regimen - single intravaginal administration of suppository. Vaginal suppositories are inserted as deeply as possible while the participant is lying down; the participant must remain in a horizontal position for 45 minutes after the administration. The total duration of volunteer participation in the study is one day. Medical observation (including gynaecological monitoring with vaginal bacterial swab test) of the subject condition after the drug administration will be carried out after 3, 6, 9, 12 and 24 hours. Repeated laboratory blood and urine tests will be performed after 24 hours. Participants of the study will be closely monitored for 24 hours after the initial administration of the drug to detect any immediate adverse events. If the subject experiences an immediate adverse event, appropriate treatment will be provided.

SUMMARY:
The study object of this clinical trial is CanProFem-AK, 100 mg suppositories. The Pharmacological group - Antifungal drug for external use. The active drug substance is the antifungal antibiotic Roseofungin 100 mg, which was developed at the "Research and Production Center of Microbiology and Virology".

According to the aims and objectives of the phase I clinical trial, the primary parameter is the study of safety and tolerability throughout the entire duration of the trial.

The phase I clinical trial of the drug CanProFem-AK 100 mg included 20 healthy female participants aged 18 to 40 years, who are on 6-12 days of their menstrual cycle. The clinical and laboratory parameters to characterize the safety of the drug: specific clinical signs and symptoms of particular importance, medical history, physical examination, biochemical analysis of blood, complete blood count with white blood cell count, and complete urine analysis.

Selection and Exclusion of Subjects: Before inclusion in a clinical trial, each participant must first sign an Informed Consent Form for Participation in the Study, followed by a screening examination, including a variety of procedures, medical history, and physical examination. Each participant in the trial will be assigned an identification number.

Study Design: open-label, single-centre, phase I clinical trial. The total duration of participation in a study is one day. The administration scheme of the drug includes the vaginal insertion of one suppository for each participant, followed by medical observation of the participants' conditions at 3, 6, 9, 12 and 24 hours after administration.

The tolerability of the drug will be assessed based on the reported participants' symptoms and sensations, and objective data obtained by the researcher during the study. The frequency and nature of adverse reactions will also be taken into account. The degree of tolerability of the study drug will be determined by three gradations: intolerance, absence of adverse drug reactions (side reactions), and adverse drug reactions (side effects) not classified as serious.

This clinical trial will be conducted following the principles formulated by the 18th World Medical Assembly (Helsinki, 1964) and the ICH guidelines for good clinical practice (GCP), as well as with all international and national laws and guidelines.

DETAILED DESCRIPTION:
The study object of this clinical trial is CanProFem-AK, 100 mg suppositories. The Pharmacological group - Antifungal drug for external use.

Fungal infections are one of the most demanding and unresolved problems of modern medicine. The number of fungal infections is growing due to the increase in the number of people with immunodeficiency diseases, oncohematological pathology, organ transplants, nursing newborns, the coronavirus pandemic, while the role of fungi that were previously considered non-pathogenic is increasing. Among fungal diseases, candidiasis, caused by fungi of the genus Candida, is of particular importance. Genital, vulvovaginal, candidiasis is a very common phenomenon. Taking into account the prevalence of candidiasis, as well as numerous cases of resistance of pathogenic fungi to drugs, an urgent task is to create new domestic effective antifungal drugs for their treatment.

Scientists from the "Research and Production Center of Microbiology and Virology" developed a new pharmaceutical antifungal drug "CanProFem-AK"® in the form of a suppository for the treatment of vaginal candidal infections. The active drug substance is the original antifungal antibiotic Roseofungin, produced by a strain of soil microorganism, that has high activity against pathogenic fungi - causative agents of human mycoses. Preclinical trials of the drug shown its safety and effectiveness in the treatment of vaginal candidiasis. The trials demonstrated that the drug exhibits high antifungal activity, therapeutic efficacy, and safety in use.

The phase I clinical trial of the drug CanProFem-AK 100 mg included 20 healthy female participants aged 18 to 40 years, who are on 6-12 days of their menstrual cycle. The clinical and laboratory parameters to characterize the safety of the drug were: specific clinical signs and symptoms of particular importance, medical history, physical examination, biochemical analysis of blood, complete blood count with white blood cell count, and complete urine analysis.

Study design: open-label, single-centre, phase I clinical trial. Dosage regimen: vaginal administration of one suppository of the studied drug (CanProFem-AK, 100 mg). The total duration of participation in a study is one day. The administration scheme of the drug includes the vaginal insertion of one suppository for each participant, followed by medical observation of the participants' conditions at 3, 6, 9, 12 and 24 hours after administration. Repeated blood and urine laboratory tests will be performed after 24 hours. Participants of the study will be closely monitored for 24 hours after the initial administration of the drug to detect any immediate adverse events. If the subject experiences an immediate adverse event, appropriate treatment will be provided.

The tolerability of the drug will be assessed based on the reported participants' symptoms and sensations, and objective data obtained by the researcher during the study. The frequency and nature of adverse reactions will also be taken into account. The degree of tolerability of the study drug will be determined by three gradations: intolerance, absence of adverse drug reactions (side reactions), and adverse drug reactions (side effects) not classified as serious.

Statistical analysis of the data is carried out based on the result of collecting the anamnestic and clinical data, as well as laboratory and instrumental research data. In addition, the volume of consultations, examinations and concomitant treatment before the study is also recorded.Data will be collected using an approved form - the Individual Registration Card.

Ethical and legal issues in clinical research: This clinical trial will be conducted following the principles established by the 18th World Medical Assembly (Helsinki, 1964) and the ICH guidelines for good clinical practice (GCP). It will be conducted in compliance with all relevant international laws and guidelines, as well as the national laws and regulations of the countries where it is conducted.

Data Collection, Record Keeping and Storage. Data collection will be conducted electronically and, to some extent, on paper.

The investigator is responsible for maintaining the confidentiality of all trial documentation, whether electronic or paper, and must implement measures to prevent accidental or premature destruction of this documentation.

All trial documentation must be retained for at least fifteen (15) years after the completion or premature termination of the clinical trial. If a longer retention period is mandated, applicable legal requirements must be taken into account.

Before destroying any important trial documents, the investigator must notify the sponsor following the completion or premature termination of the clinical trial.

Financing and insurance. All financing and insurance matters will be outlined in the agreement between the Sponsor and the Contractor.

Publications. Investigator agrees not to publish or disclose the study and/or its results without prior written permission from the study sponsor, provided that the sponsor will not withhold such permission without a valid reason. The researcher will not use the sponsor's name in any advertising materials or publications without the sponsor's prior written consent. Likewise, the sponsor will not use the investigator's or their staff's names in advertising materials or publications without first obtaining their written consent. The sponsor retains the right to publish the study results at any time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers aged 18-40 years with verified health status and no chronic or acute systemic or dermatological diseases.
* Willingness to voluntarily participate in the study.

Exclusion Criteria:

* Individuals with chronic diseases (tuberculosis, hepatitis, HIV infection, diabetes mellitus, cancer), chronic renal failure, chronic liver failure, exacerbations of chronic diseases;
* Individuals participating in parallel clinical trials of other drugs, or who participated within 3 months from the start of the current study;
* Individuals from the category of "vulnerable patients" (homeless, military personnel, incapacitated persons, patients in emergency situations, and other individuals who may be the subject of pressure);
* Patients with an allergy in their medical history and during screening (medicinal, pollen and other types);
* Patients with a history of oncopathology or a family history of oncopathology (the presence of oncopathology among close relatives);
* Patients with hypersensitivity to one of the components of the study drug;
* Pregnancy and breastfeeding;
* Patient's refusal to perform the procedures required by the protocol and inability to adhere to the procedure schedule.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
General indicators for safety evaluation of a studied drug: | 24 hours
  * Absence of allergic reactions and clinically significant changes in blood count
  * Analysis of biochemical blood test indicators
  * Complete blood count with white blood cell count, and complete urine analysis
  * Absence of changes in the general somatic condition of volunteers during the study period (physical examination). Absence of side effects.
Tolerability of the studied drug | 24 hours
  The degree of tolerability of the studied drug will be determined by three gradations:
  * Intolerance: The appearance of local signs of allergy/pseudoallergy and systemic signs, such as tachycardia (heart rate over 90 per minute for 30 minutes after administration), decreased blood pressure (less than 100/60 mm Hg for 30 minutes after application), or serious adverse drug reactions.
  * Absence of adverse drug reactions (side effects).
  * Adverse drug reactions (side effects) not classified as serious.

CONTACTS AND LOCATIONS:
Locations (1):
- MIPO Clinic LLP, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ongarbayeva N., Balgimbayeva А., Baimakhanova B., Sadanov А., Lakhk O., Orazymbet S., Trenozhnikova L., Berezin V., Bogoyavlenskiy A. Pharmacotherapy for vulvovaginal candidiasis // Microbiology and Virology. - 2024. - 2(45). - pp. 83-107. https://doi.org/10.53729/MV-AS.2024.02.06
- [Background] Sadanov A.K., Ibragimova L.N., Balgimbayeva A.S., Trenozhnikova L.P., Tugelbay G.E., Berezin V.E., Turlybaeva Z.Zh. Suppositories with antifungal and antiviral activity. - Utility patent No. 5056 dated 10/09/2020.
- [Background] Certificate for the Trademark "КанПроФем-АК/CanProFem-AK", No. 69692 dated July 30, 2020.